CLINICAL TRIAL: NCT00002784
Title: Randomized Trial of High-dose Epirubicin and Cyclophosphamide x 3 Supported by Peripheral Blood Progenitor Cells Versus Anthracycline and Cyclophosphamide x 4 Followed by Cyclophosphamide, Methotrexate, and 5-fluorouracil x 3 as Adjuvant Treatment for High Risk Operable Stage ii and Stage Iii Breast Cancer in Premenopausal and Young Postmenopausal (Less Than or Equal to 65 Yrs) Patients.
Brief Title: High-Dose Combination Chemotherapy Plus Peripheral Stem Cell Transplantation Compared With Standard Combination Chemotherapy in Treating Women With High-Risk Breast Cancer
Acronym: 15-95
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064834; IBCSG-15-95; EU-96021
Record Dates: First submitted 1999-11-01; First posted 2004-07-29 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; CMF regimen; Cyclophosphamide; Doxorubicin; Epirubicin; Fluorouracil; Mesna; Methotrexate; Tamoxifen; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard chemotherapy (Active Comparator): EC/AC x 4 followed by CMF x 3 and tamoxifen to 5 years after randomization.
  Interventions: Drug: CMF regimen; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: epirubicin hydrochloride; Drug: fluorouracil; Drug: methotrexate; Drug: tamoxifen citrate; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy
- Dose-intensive EC (Experimental): High-dose EC x 3 supported by peripheral blood progenitor cells and tamoxifen to 5 years after randomization.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: mesna; Drug: tamoxifen citrate; Procedure: peripheral blood stem cell transplantation; Radiation: low-LET electron therapy; Radiation: low-LET photon therapy

INTERVENTIONS:
Biological: filgrastim — Filgrastim 10 mg/kg/d sc for 6 days after randomization.
  Arms: Dose-intensive EC
Drug: CMF regimen — Cyclophosphamide 100 mg/m2 orally days 1 - 14, methotrexate 40 mg/m2 iv days 1 and 8, 5-fluorouracil 600 mg/m2 iv days 1 and 8. Repeat every 28 days.
  Arms: Standard chemotherapy
Drug: cyclophosphamide — For high-dose EC arm: cyclophosphamide 4 gm/m2 iv as 4 divided doses. For standard chemotherapy arm: cyclophosphamide 600 mg/m2 iv day 1 of 21-day EC cycles, and cyclophosphamide 100 mg/m2 orally on days 1-14 of 28-day CMF cycles.
Drug: doxorubicin hydrochloride — Doxorubicin 60 mg/m2 iv on day 1 of 21-day cycles of AC.
  Arms: Standard chemotherapy
Drug: epirubicin hydrochloride — Epirubicin 90 mg/m2 iv on day 1 of 21-day cycles of EC.
  Arms: Standard chemotherapy
Drug: fluorouracil — 5-fluorouracil 600 mg/m2 iv days 1 and 8 of 28-day cycles of CMF.
  Arms: Standard chemotherapy
Drug: mesna — MESNA (7.2 gm/m2) on days 2 and 3 of 21-day cycles of dose-intensive EC.
  Arms: Dose-intensive EC
Drug: methotrexate — Methotrexate 40 mg/m2 iv on days 1 and 8 of 28-day cycles of CMF.
  Arms: Standard chemotherapy
Drug: tamoxifen citrate — Tamoxifen 20mg daily for 5 years or until relapse.
Procedure: peripheral blood stem cell transplantation — Peripheral blood progenitor cells (PBPC) infusion on day 5 of each 21-day cycle of dose-intensive EC.
  Arms: Dose-intensive EC
Radiation: low-LET electron therapy — Radiation therapy to the conserved breast is mandatory, to be carried out according to the prospectively defined guidelines of each participating institution; either after all chemotherapy or integrated into CMF as agreed per institution. Radiotherapy to the chest wall following mastectomy is optional according to the prospectively defined guidelines of each participating institution.
Radiation: low-LET photon therapy — radiation therapy to the conserved breast is mandatory, to be carried out according to the prospectively defined guidelines of each participating institution; either after all chemotherapy or integrated into CMF as agreed per institution. Radiotherapy to the chest wall following mastectomy is optional according to the prospectively defined guidelines of each participating institution.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. It is not yet known if high-dose combination chemotherapy plus peripheral stem cell transplantation is more effective than standard combination chemotherapy for breast cancer.

PURPOSE: Randomized phase III trial to compare high-dose combination chemotherapy plus peripheral stem cell transplantation with standard combination chemotherapy in treating women with stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the survival, disease-free survival, and systemic disease-free survival of women with high-risk, operable stage II/III breast cancer treated with three courses of dose-intensive epirubicin/cyclophosphamide (EC) supported by granulocyte colony-stimulating factor (G-CSF) and G-CSF-mobilized peripheral blood stem cells vs. standard EC followed by cyclophosphamide/methotrexate/fluorouracil. II. Compare the toxicity, duration of quality-adjusted time without symptoms and toxicity, and quality of life associated with these two treatments. III. Evaluate the cost effectiveness of these two treatments.

OUTLINE: This is a randomized study. Patients are stratified by estrogen receptor status and menopausal status. Within 6 weeks of surgery, patients in the first group receive epirubicin (preferred) or doxorubicin plus cyclophosphamide every 3 weeks for 4 courses followed by conventional cyclophosphamide, methotrexate, and fluorouracil (CMF) every 4 weeks for 3 courses. Patients in the second group undergo stem cell mobilization and harvest with granulocyte colony-stimulating factor (G-CSF) followed within 10 weeks of surgery by high-dose chemotherapy with epirubicin and cyclophosphamide followed by peripheral blood stem cell rescue and G-CSF. All patients receive adjuvant tamoxifen, and patients who underwent lumpectomy prior to entry are required to receive adjuvant radiotherapy (radiotherapy is optional for patients who underwent mastectomy prior to entry). Patients are followed every 3 months for 2 years, then q 6 months for 3 years, then yearly.

PROJECTED ACCRUAL: 210 patients will be accrued over 4 years to provide 195 evaluable patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven breast carcinoma in one of the following categories: 10 or more involved axillary nodes 5 or more involved axillary nodes and either: Primary tumor estrogen receptor (ER)-negative (less than 10 femtomoles per milligram of cytosol protein) T3 tumor (regardless of ER status) Total mastectomy or breast-conserving procedure (lumpectomy or quadrantectomy) required within 6 weeks prior to randomization Tumor confined to breast and axillary nodes (T1a-c, T2, or T3, N1-2, M0 by the UICC staging system) The following conditions exclude entry: Satellite skin nodules distant from the primary tumor Supraclavicular node involvement Inoperable, matted axillary nodes Fixation of primary tumor to chest wall (excluding pectoralis major) Bilateral breast cancer (any mass in opposite breast unless biopsy-proven benign) Hot spots on bone scintigram (unless confirmed to be benign) Skeletal pain of unknown cause Hormone receptor status: ER status determination preferred, but not required

PATIENT CHARACTERISTICS: Age: 16-65 Sex: Women only Menopausal status: Any status Performance status: ECOG 0-2 Hematopoietic: WBC at least 4,000 Platelets at least 100,000 Hepatic: Bilirubin no greater than 1.1 mg/dL (20 micromoles/L) AST no greater than twice normal Renal: Creatinine no greater than 1.3 mg/dL (120 micromoles/L) Cardiovascular: Left ventricular ejection fraction greater than 50% by MUGA Other: No second malignancy except: Basal cell carcinoma Adequately treated carcinoma in situ of the cervix No significant nonmalignant disease that would preclude participation No psychiatric or addictive disorder that would compromise informed consent or participation No pregnant or nursing women Adequate contraception strongly advised for fertile women

PRIOR CONCURRENT THERAPY: No prior therapy for breast cancer other than surgery (see Disease Characteristics)

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 1996-06; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Disease-free survival. | 16 years after randomization.
  Time from randomization to recurrence (including recurrence isolated to the breast), metastasis, appearance of a second primary tumor, or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival. | 16 years after randomization.
  Time from randomization to death from any cause.
Toxicity. | 5 years after randomization.
  Morbidity information was recorded using standard toxicity criteria.
Quality of life. | 16 years after randomization.
  Quality of life was assessed using standard International Breast Cancer Study Group instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Basser, MD, Study Chair — Melbourne Health
Locations (11):
- Australia (5):
  - Newcastle Mater Misericordiae Hospital, Newcastle, New South Wales
  - Royal Prince Alfred Hospital, Sydney, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
- Switzerland (6):
  - Swiss Institute for Applied Cancer Research, Bern
  - Inselspital, Bern, Bern
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Istituto Oncologico della Svizzera Italiana, Lugano
  - Kantonsspital - Saint Gallen, Sankt Gallen
  - Universitaetsspital, Zurich

REFERENCES:
- [Background] Pestalozzi BC, Zahrieh D, Mallon E, Gusterson BA, Price KN, Gelber RD, Holmberg SB, Lindtner J, Snyder R, Thurlimann B, Murray E, Viale G, Castiglione-Gertsch M, Coates AS, Goldhirsch A; International Breast Cancer Study Group. Distinct clinical and prognostic features of infiltrating lobular carcinoma of the breast: combined results of 15 International Breast Cancer Study Group clinical trials. J Clin Oncol. 2008 Jun 20;26(18):3006-14. doi: 10.1200/JCO.2007.14.9336. Epub 2008 May 5. PMID 18458044
- [Background] Keshaviah A, Dellapasqua S, Rotmensz N, Lindtner J, Crivellari D, Collins J, Colleoni M, Thurlimann B, Mendiola C, Aebi S, Price KN, Pagani O, Simoncini E, Castiglione Gertsch M, Gelber RD, Coates AS, Goldhirsch A. CA15-3 and alkaline phosphatase as predictors for breast cancer recurrence: a combined analysis of seven International Breast Cancer Study Group trials. Ann Oncol. 2007 Apr;18(4):701-8. doi: 10.1093/annonc/mdl492. Epub 2007 Jan 20. PMID 17237474
- [Result] Colleoni M, Sun Z, Martinelli G, Basser RL, Coates AS, Gelber RD, Green MD, Peccatori F, Cinieri S, Aebi S, Viale G, Price KN, Goldhirsch A; International Breast Cancer Study Group. The effect of endocrine responsiveness on high-risk breast cancer treated with dose-intensive chemotherapy: results of International Breast Cancer Study Group Trial 15-95 after prolonged follow-up. Ann Oncol. 2009 Aug;20(8):1344-51. doi: 10.1093/annonc/mdp024. Epub 2009 May 25. PMID 19468030
- [Result] International Breast Cancer Study Group; Basser RL, O'Neill A, Martinelli G, Green MD, Peccatori F, Cinieri S, Coates AS, Gelber RD, Aebi S, Castiglione-Gertsch M, Viale G, Price KN, Goldhirsch A. Multicycle dose-intensive chemotherapy for women with high-risk primary breast cancer: results of International Breast Cancer Study Group Trial 15-95. J Clin Oncol. 2006 Jan 20;24(3):370-8. doi: 10.1200/JCO.2005.03.5196. PMID 16421418
- [Result] Basser RL, Abraham R, To LB, Fox RM, Green MD. Cardiac effects of high-dose epirubicin and cyclophosphamide in women with poor prognosis breast cancer. Ann Oncol. 1999 Jan;10(1):53-8. doi: 10.1023/a:1008390203340. PMID 10076722
- [Result] Basser RL, To LB, Collins JP, Begley CG, Keefe D, Cebon J, Bashford J, Durrant S, Szer J, Kotasek D, Juttner CA, Russell I, Maher DW, Olver I, Sheridan WP, Fox RM, Green MD. Multicycle high-dose chemotherapy and filgrastim-mobilized peripheral-blood progenitor cells in women with high-risk stage II or III breast cancer: five-year follow-up. J Clin Oncol. 1999 Jan;17(1):82-92. doi: 10.1200/JCO.1999.17.1.82. PMID 10458221
- [Result] Basser RL, To LB, Begley CG, Juttner CA, Maher DW, Szer J, Cebon J, Collins JP, Russell I, Olver I, et al. Adjuvant treatment of high-risk breast cancer using multicycle high-dose chemotherapy and filgrastim-mobilized peripheral blood progenitor cells. Clin Cancer Res. 1995 Jul;1(7):715-21. PMID 9816037